CLINICAL TRIAL: NCT07233213
Title: An Open-label, Single-arm, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of Human Immunoglobulin for Intravenous Injection (5%) in the Treatment of Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: An Open-label Study of Intravenous Immunoglobulin (5%) for the Treatment of Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grand Shuyang Life Sciences (Chengdu) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLS-IVIG-A01-III
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: autoimmune hemorrhagic disease; hemorrhage
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Hemorrhage | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, open-label, multicenter phase III clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who meet all of the following criteria are eligible to be included in this clinical trial. (Experimental): Investigational Product Name: Human immunoglobulin (pH4) for intravenous injection Formulation: Injection Specification: 5 g/vial (5%, 100 mL) Manufacturer: Grand Shuyang Life Sciences (Chengdu) Co., Ltd. Administration: Direct intravenous drip at the initial rate of 1.0 ml/min (about 20 drops/min). If there is no adverse reaction after 15 minutes, it can be gradually increased. The fastest drip rate should not exceed 3.0 ml/min (about 60 drops/min).
  Dosage: Direct intravenous drip, 0.4 g/kg daily for 5 consecutive days. The body weight value is kept as an integer (rounded off), and the dose calculated by body weight is within the allowable range of the theoretical dose ± 5 ml. For example, if the body weight of a patient is 57 kg and the theoretical dosage is 22.8 g/day based on 0.4 g/kg per day of human immunoglobulin for intravenous injection (5%, 5g/100ml strength), 456 ml of drug will be required, so the actual dose ranging from 451 ml to 461 ml is allowable.
  Interventions: Drug: Human immunoglobulin (pH4) for intravenous injection

INTERVENTIONS:
Drug: Human immunoglobulin (pH4) for intravenous injection — Administration: Direct intravenous drip at the initial rate of 1.0 ml/min (about 20 drops/min). If there is no adverse reaction after 15 minutes, it can be gradually increased. The fastest drip rate should not exceed 3.0 ml/min (about 60 drops/min).
  Direct intravenous drip, 0.4 g/kg daily for 5 consecutive days. The body weight value is kept as an integer (rounded off), and the dose calculated by body weight is within the allowable range of the theoretical dose ± 5 ml. For example, if the body weight of a patient is 57 kg and the theoretical dosage is 22.8 g/day based on 0.4 g/kg per day of human immunoglobulin for intravenous injection (5%, 5g/100ml strength), 456 ml of drug will be required, so the actual dose ranging from 451 ml to 461 ml is allowable.

SUMMARY:
It is a clinical trial of a medicinal product Human Immunoglobulin for Intravenous Injection (5%) manufactured by Grand Shuyang Life Sciences (Chengdu) Co., Ltd. (hereinafter referred to as 5% IVIG). This clinical study is conducted to evaluate the efficacy and safety of 5% IVIG in patients with primary Immune Thrombocytopenia (ITP).

The study includes 4 periods and 9 visits (designated as V):

* Screening period (V1: 14 days before the first administration, preliminary examination);
* Baseline Period (V2: within 24 h before the first dose, Day 0);
* Treatment Period (V3: Day 1 to Day 5, administration of the drug in a hospital setting);
* Follow-up Period (V4-V9: visits to Study Site on Day 6, Day 7, Day 14 + 2, Day 21 + 3, Day 28 + 4, and Day 90 (+ 14) after the first dose).

In this study, the investigational product 5% IVIG will be administered at a dose of 0.4 g/kg/day (direct intravenous drip) for 5 consecutive days. The total duration of your participation in the study will be approximately 104 days. The investigational product will only be provided during the study period. It will not be supplied after the study ends.

The study will be conducted at clinical centers in Turkey. It is planned to obtain data from 36 patients included in the study (no more than 48 screened patients).

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form, male or female patients aged ≥ 18 years and ≤ 65 years;
2. Patients with clinically confirmed chronic ITP (i.e., the course of disease > 12 months from diagnosis to signing the informed consent form);
3. Patients who did not use glucocorticoids for at least 2 weeks before the first dose or used a maintenance dose of glucocorticoids for at least 2 weeks before the first dose, and did not plan to increase the dosage of glucocorticoids or add other platelet-elevating drugs within 4 weeks after the first dose;
4. Platelet count < 30 × 109/L;
5. Patients who understand the procedures and methods of this study, are willing to sign the informed consent form and complete the study in strict accordance with the clinical study protocol.

Exclusion Criteria:

1. Patients who are known or suspected to be allergic to human immunoglobulin or other plasma proteins and/or blood products, as well as excipients of the investigational drug, including those with a history of steroid hormone allergy;
2. BMI ≥ 30 kg/m2;
3. Secondary thrombocytopenia;
4. Patients with the following clinical manifestations or disease history at screening:

   * Hemoglobin <90 g/L or combined with immune hemolytic anemia;

     * Chronic or recurrent neutropenia (defined as absolute neutrophil count < 1.5 × 109/L);

       * Patients with abnormal liver function: defined as ALT and/or AST > 3 times of the upper limit of normal; and/or total bilirubin ≥ 1.5 times of the upper limit of normal;

         * Patients with related diseases of renal impairment, or serum creatinine ≥ 1.5 times the upper limit of normal value or creatinine clearance < 60 mL/min; ⑤. Patients with dysglycemia, including: Confirmed diagnosis of type 1/2 diabetes mellitus with HbA1c ≥7.0%, Fasting glucose ≥7.0 mmol/L (126 mg/dL), or Random glucose ≥11.1 mmol/L (200 mg/dL);

           ⑥. Blood diseases with coagulation factor defects;

           ⑦. Selective IgA deficiency patients with anti-IgA antibodies;

           ⑧. Patients with uncontrollable hypertension (SBP>160 mmHg or DBP>100 mmHg) or hypotension (SBP<90 mmHg or DBP<60 mmHg);

           ⑨. Patients with hyperviscosity, severe cardiovascular and cerebrovascular diseases (such as TIA, stroke, thrombotic disease, congestive heart failure of NYHA classification III/IV, arrhythmia requiring drug therapy (unstable angina pectoris) or myocardial infarction, etc.) and other serious systemic diseases before signing the informed consent form, who are not suitable for enrollment as judged by the investigator;

           ⑩. Suffering from mental illness, obvious mental disorder or epilepsy; incapacitated or cognitively impaired;
5. Patients who failed to respond to previous treatment with human immunoglobulin for intravenous injection or anti-D human immunoglobulin;
6. Patients who had received treatment with human immunoglobulin for intravenous injection or anti-D human immunoglobulin within 4 weeks prior to the first dose, or any other treatment with blood, blood products or blood derivatives within 4 weeks before signing the informed consent form;
7. Patients who have received recombinant human thrombopoietin or eltrombopag and other receptor agonists within 2 weeks prior to the first dose (except for those who are ineffective after stable treatment > 2 weeks), or other drugs with clear indications of increasing platelet count;
8. Patients who have received immunosuppressive or other immunomodulatory drugs within 3 weeks prior to the first dose (except for the following cases: glucocorticoids with stable dose and no dose change for > 2 weeks, and patients who failed to respond to stable treatment with azathioprine, cyclophosphamide or danazol for > 12 weeks);
9. Patients who received rituximab within 8 weeks prior to the first dose;
10. Patients who have been vaccinated with live attenuated vaccines within 8 weeks prior to the first dose or are planned to be vaccinated during the trial treatment, such as poliomyelitis vaccine, measles vaccine, rubella vaccine, mumps vaccine and varicella virus vaccine; patients who are planned to be vaccinated with measles vaccine within 1 year after the administration of the investigational drug;
11. Patients scheduled for surgery during the trial and requiring transfusion of blood or blood products;
12. Those who planned to continue taking non-steroidal anti-inflammatory drugs, warfarin and other drugs that affect platelet aggregation or coagulation function due to medical history during the trial;
13. Patients who tested positive for any of HBs antigen (or nucleic acid test), HCV antibody (or nucleic acid test), Treponema pallidum antibody and HIV antibody (or nucleic acid test) at screening;
14. Acute bacterial or acute viral infections that still require antibiotic treatment after enrollment;
15. Pregnant and lactating women who have aborted for less than 30 days before signing the informed consent form (currently breastfeeding or currently not artificially breastfeeding but less than one year after delivery); female patients or spouses of male patients who plan to get pregnant or donate eggs or male patients who donate sperm during the trial and within 90 days after the last dose, and effective contraception cannot be guaranteed;
16. Patients with a history of drug abuse or drug addiction;
17. Patients who have participated (already included) in clinical trials of other drugs or medical devices within 3 months before signing the informed consent form;
18. The survival time is expected to be less than 3 months, or the patients with other concomitant diseases are severely ill and may be dying during the treatment period and follow-up period. In the investigator's opinion, the efficacy cannot be evaluated or it is unlikely to complete the expected course of treatment and follow-up;
19. Patients with poor compliance or who are not suitable to participate in this trial for other reasons as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Improved platelet response within 7 days of the first transfusion | Within 7 days of the first transfusion
  The response rate is defined as the proportion of patients whose platelet count > 30 × 109/L and increased to more than 2 times of baseline within 7 days after the first IVIg transfusion and absence of bleeding.

SECONDARY OUTCOMES:
Time to and duration (days) of platelet count > 30 × 109/L | Within 7 days after the first IVIg infusion
  Time to and duration (days) of platelet count > 30 × 109/L and increased to more than 2-fold baseline within 7 days after the first IVIg infusion without bleeding
Peak and time to peak platelet count | After the first infusion of IVIg
  Peak and time to peak platelet count after the first infusion of IVIg (days)
Number and percentage of patients achieving complete response (CR), response (R), non-response (NR) and relapse | Within 28 days after the first infusion
  Number and percentage of patients achieving complete response (CR), response (R), non-response (NR) and relapse within 28 days after the first infusion
Time to arrival of CR or R response and duration of response | Within 28 days after the first infusion
  Time to arrival of CR or R response and duration of response within 28 days after the first infusion
Effective rate | On the 14th, 21st and 28th day after the first dose
  Effective rate on the 14th, 21st and 28th day after the first dose
ITP bleeding scale score of patients | Within 7 days after the first infusion, and on Days 14, 21 and 28
  ITP bleeding scale score of patients within 7 days after the first infusion, and on Days 14, 21 and 28
ITP bleeding scale score | On Day 7 after the first dose of treatment
  ITP bleeding scale score on Day 7 after the first dose of treatment for all bleeding events during follow-up

CONTACTS AND LOCATIONS:
Locations (9):
- Turkey (Türkiye) (9):
  - Hacettepe University Faculty of Medicine, Ankara, Altındağ
  - İnönü University Turgut Ozal Medical Center Training and Research Hospital, Malatya, Battalgazi
  - İstanbul University, Istanbul Faculty of Medicine, Istanbul, Fatih
  - Erciyes University Hematology Hospital, Kayseri, Melikgazi
  - VM Medical Park Mersin, Mersin, Mezitli
  - Antalya Training and Research Hospital, Antalya, Muratpaşa
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Eğitim ve Araştırma Hastanesi, Ankara, Yenimahalle
  - Adana City Education and Research Hospital, Hematology Department, Adana, Yüreğir
  - Gaziantep University Şahinbey Training and Research Hospital, Gaziantep, Şehitkamil